CLINICAL TRIAL: NCT06523998
Title: Retrospective Descriptive Observational Study of the Epidemiological, Clinical and Therapeutic Profile of Patients With Rare Infections of Dermatological Interest at Three Major Reference Hospitals in Costa Rica From 2019-2023
Brief Title: A Study on Rare Dermatological Infections Conducted at Three Major Reference Hospitals in Costa Rica.
Status: Completed | Type: Observational
Sponsor: Caja Costarricense de Seguro Social (Other Government)
Responsible Party: Principal Investigator, Daniel Barquero Orias, Medical Doctor, Caja Costarricense de Seguro Social
Other Study IDs: R023-SABI-00344
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Sporotrichosis; Chromomycosis; Actinomycosis; Nocardiosis; Mycetoma; Mycobacterial Cutaneous Infection; Coccidioidomycosis; Blastomycosis; Paracoccidioidomycosis; Phaeomycosis
Keywords: Bacterial Infections and Mycoses; Infectious Skin Diseases; Sporotrichosis; Chromoblastomycosis; Mycetoma; Non-tuberculous mycobacteria
MeSH Terms: conditions — Sporotrichosis; Chromoblastomycosis; Actinomycosis; Nocardia Infections; Mycetoma; Coccidioidomycosis; Blastomycosis; Paracoccidioidomycosis; Phaeohyphomycosis; Bacterial Infections and Mycoses; Skin Diseases, Infectious

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Costa Rica there are some descriptive studies of some of these rare infectious diseases (sporotrichosis, chromomycosis and mycetomas); however, there are no recent published reports. Most of the publications on the subject date back to the previous century; from 2000 to the present year there are only publications of small series of cases, so the current behavior of these skin infections is unknown. The primary objective is to analyze the epidemiological, clinical, and therapeutic profile and determine the risk factors in patients with a diagnosis of rare infections of dermatological interest treated at Hospital México, Hospital Rafael Calderón Guardia, and Hospital San Juan de Dios during the period 2019-2023.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years, regardless of gender and ethnic group.
2. Patients who during the period from January 1, 2019 to December 31, 2023 received medical care at the Hospital Rafael Ángel Calderón Guardia, Hospital México and Hospital San Juan de Dios.
3. Subjects who meet a confirmed microbiological, histological and/or molecular diagnosis of sporotrichosis, chromomycosis, actinomycosis, nocardiosis, mycetoma, mycobacterial infection, coccidioidomycosis, blastomycosis, paracoccidioidomycosis, cutaneous nocardiosis and pheomycotic abscess (either through the unique digital health record, pathology registries, clinical laboratory service database of each hospital, clinical laboratory of the University of Costa Rica and Instituto Costarricense de Investigación y Enseñanza en Nutrición y Salud).
4. Subjects diagnosed at a private level and referred to continue medical care at Hospital Rafael Ángel Calderón Guardia, Hospital México and Hospital San Juan de Dios.

Exclusion Criteria:

1. The research team may exclude patients who have an unconfirmed diagnosis, an erroneous diagnosis, or have participated in the study before, as they may hinder the ability to obtain satisfactory data to achieve the study's objectives.
2. Patients who have more than 30% of the variables required for analysis missing will also be excluded from the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years with confirmed microbiological, histological and/or molecular diagnosis of sporotrichosis, chromomycosis, actinomycosis, nocardiosis, mycetoma, mycobacterial infection, coccidioidomycosis, blastomycosis, paracoccidioidomycosis, cutaneous nocardiosis and pheomycotic abscess diagnosed and/or treated at Hospital México, Hospital Rafael Calderón Guardia, and Hospital San Juan de Dios during the period 2019-2023.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Analyze epidemiological, clinical, and therapeutic profile | 5 year
  Analyze the epidemiological, clinical, and therapeutic profile and determine the risk factors in patients with a diagnosis of rare infections of dermatological interest treated at Hospital México, Hospital Rafael Calderón Guardia, and Hospital San Juan de Dios during the period 2019-2023.
Determine the risk factors | 5 year
  Analyze the epidemiological, clinical, and therapeutic profile and determine the risk factors in patients with a diagnosis of rare infections of dermatological interest treated at Hospital México, Hospital Rafael Calderón Guardia, and Hospital San Juan de Dios during the period 2019-2023.
Determine the diagnostic methods | 5 year
  Determine the diagnostic methods utilized for each case, including culture, histological techniques, and molecular testing.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Barquero Orias, MD, Principal Investigator — Caja Costarricense de Seguro Social
Locations (3):
- Costa Rica (3):
  - Hospital Rafael Ángel Calderón Guardia, San José
  - Hospital San Juan de Dios, San José
  - Hospital México, San José

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolognia JL, Schaffer JV, Cerroni L, Callen JP. Dermatología. 4th ed. Barcelona: Elsevier; 2019.
- [Background] Kang S, Amagai M, Bruckner AL, Enk AH, Margolis DJ, McMichael AJ, et al. Fitzpatrick's Dermatology. 9th ed. New York: McGraw-Hill Education; 2019.
- [Background] Trejos A. La cromoblastomicosis como problema micológico [Tesis de grado para optar por el título de licenciatura en Microbiología]. San José, Costa Rica: Universidad de Costa Rica, 1954.
- [Background] Trejos A. Cladosporium carrionii n. sp. and the problem of Cladosporia isolated from chromoblastomycosis. Rev Biol Trop. 1954, 2(1):75-112.
- [Background] Mora M, Molina B, Moya A. Cromoblastomicosis por Cladophialophora Carrionnii: Primer caso descrito en literatura costarricense. Rev. méd. Costa Rica Centroam. 2010;67(594):373-6.
- [Background] Romero A, Trejos A. La cromomicosis en Costa Rica. Rev Biol Trop. 1953;1(2):95-115.
- [Background] Soto L, Jaikel D. Cromoblastomicosis: Situación en Costa Rica. Rev. méd. Costa Rica Centroam. 2014;71(613):737-44.
- [Background] Salazar K. Esporotricosis y cromoblastomicosis en San Ramón de Costa Rica. Acta Med Costarr. 2022;64(3):1-5. Disponible en https://doi.org/10.51481/amc.v64i3.1224
- [Background] Solano E. Cromomicosis. Acta Med Costarr. 1966;9(2):77-85.
- [Background] Astorga E, Bonilla E, Martínez C, Mora W. Cromomicosis (Nuevos casos de Cromomicosis tratados con Anfotericina B y 5·Fluorcitosina en forma simultánea). Rev. Méd. de Costa Rica. 1980;47(479):17-22.
- [Background] Sáenz L, Morera P. Sobre un caso de blastomicosis suramericana asociada a cromomicosis. Acta Med Costarr. 1963;6(1):55-71.
- [Background] Alice E. Ecología de Sporothrix schenkii. Rev Méd de Costa Rica. 1982;49(479):81-6.
- [Background] Rodríguez J. Aspectos clínicos, epidemiológicos y ecológicos sobre 100 casos de Esporotricosis en Costa Rica. Revista costarricense de Ciencias Médicas. 1992;12:29-36.
- [Background] González J, Rodríguez J. Tres casos de Esporotricosis. Revista costarricense de Ciencias Médicas. 1990;12:57-9.
- [Background] Jaramillo O. Esporotricosis en Costa Rica: Estudio clínico epidemiológico y terapéutico de cien casos. Boletín Médico del Seguro Social de Costa Rica. 1972;1(4):27-37.
- [Background] Rodríguez J, Gamboa A, Alvarado F. Etiología y epidemiología de los micetomas en Costa Rica. Rev. iberoamer. micol. 1988;5:144-8.
- [Background] Trejos A, Romero A. Contribución al estudio de las blastomicosis en Costa Rica. Rev Biol Trop. 1953;1(1):63-81.
- [Background] Astorga E, Mora W, Rodríguez A. Tratamiento de la Paracoccidioidomicosis con Ketoconazol (Primer caso en Costa Rica). Rev. Méd. de Costa Rica. 1986;53(494):1-3.
- [Background] Fernández K, Quirós JL. Paracoccidiodomicosis: (Reporte de siete casos). Rev. méd. Costa Rica Centroam. 2008;65(582):41-7.
- [Background] Kawer A, Madrigal L, Mata F. Paracoccidioidomicosis en lengua. Rev. méd. Costa Rica Centroam. 2011;68(599):505-8.
- [Background] Bonilla E, Miranda M, Mata L. Reporte del primer caso de Nocardiasis en Costa Rica. Acta Med Costarr. 1960;3(1):51-5.
- [Background] Cueva A. Nocardiosis. Acta Med Costarr. 1968;11(1):45-51. 23.
- [Background] CASTRO A, TREJOS A. [Confirmation of the first Central American cas of coccidioidomycosis]. Rev Med Costa Rica. 1951 Apr;18(204):89-90. No abstract available. Undetermined Language. PMID 14854495
- [Background] Hidalgo W, Xinirachs H, Cappella E, Solano E. Un caso de actinomicosis cervicofacial por Actinomyces bovis. Rev Biol Trop. 1960;8(2):155-63.
- [Background] Hidalgo W, Morera P, Hernández VM, Suárez A, Céspedes R. Criptococosis Estudio del primer caso confirmado en Costa Rica. Acta Med Costarr. 1960;3(5):221-35.
- [Background] Brizuela S, Montero N. Criptococosis asociado a VIH/SIDA (A propósito de un paciente). Rev. méd. Costa Rica Centroam. 2013;70(605):43-7.
- [Background] Mora J, Salazar J, Calderón C, García R. Rinosporidiosis en Costa Rica. (Revisión del tema e informe del primer caso en nuestro país). Acta Med Costarr. 1985;28(2):122-5.
- [Background] Riggioni S, Díaz S. Lacaziosis: Micosis cutánea profunda, Reporte de un caso. Rev. clín. esc. med. UCR-HSJD. 2015 Jun 29;5(3). https://doi.org/10.15517/rc_ucr-hsjd.v5i3.19916